CLINICAL TRIAL: NCT04784559
Title: A Phase 3, Multicentre, Randomised, Controlled Trial to Determine the Efficacy and Safety of Two Dose Levels of Plitidepsin Versus Control in Adult Patient Requiring Hospitalisation for Management of Moderate COVID-19 Infection
Brief Title: Trial to Determine the Efficacy/Safety of Plitidepsin vs Control in Patients With Moderate COVID-19 Infection
Acronym: Neptuno
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor has decided to end the study prematurely based on significant difficulties in the recruitment of patients, despite the implementation of corrective measures that still failed to increase the accrual rate required for a feasible completion.
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL-D-003-20; 2020-005951-19 (EudraCT Number)
Record Dates: First submitted 2021-03-04; First posted 2021-03-05 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — plitidepsin; Dexamethasone; remdesivir; favipiravir

STUDY DESIGN:
Intervention Model Description: Patients Will be randomised in 1:1:1 to: Plitidepsin 1.5 mg arm, Plitidepsin 2.5 mg arm and Control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plitidepsin 1.5 mg arm (Experimental): Patients will receive plitidepsin 1.5 mg/day intravenous (IV) in addition to dexamethasone on days 1 to 3.
  Interventions: Drug: Plitidepsin; Drug: Dexamethasone
- Plitidepsin 2.5 mg arm (Experimental): Patients will receive plitidepsin 2.5 mg/day IV in addition to dexamethasone on days 1 to 3.
  Interventions: Drug: Plitidepsin; Drug: Dexamethasone
- Control arm (Active Comparator): Patients will receive dexamethasone IV on Days 1 to 3. Additionally, in accordance with local treatment guidelines, patients in this group may receive a regulatory-approved antiviral treatment.
  Interventions: Drug: Dexamethasone; Drug: Remdesivir; Drug: Favipiravir

INTERVENTIONS:
Drug: Plitidepsin — Plitidepsin 2 mg powder is provided as a sterile, preservative-free, and white to off-white lyophilised powder/cake comprising 2 mg plitidepsin and mannitol in a single-dose, 10 mL clear type 1 glass vial.
  Solvent for plitidepsin is provided as a sterile, preservative-free, clear, slightly viscous aqueous liquid (4 mL) containing macrogolglycerol ricinoleate and ethanol in a single-dose type 1 clear glass ampoule.
  For administration, vial contents are reconstituted by addition of 4 mL of solvent for plitidepsin to obtain a slightly yellowish solution containing 0.5 mg/mL plitidepsin with mannitol, macrogolglycerol ricinoleate and ethanol excipients. The required amount of plitidepsin reconstituted solution is added to bag containing 0.9% sodium chloride or 5% glucose for IV injection and administered as an IV infusion over 60 minutes.
  Arms: Plitidepsin 1.5 mg arm; Plitidepsin 2.5 mg arm
Drug: Dexamethasone — Detailed information about the formulation, posology, packaging and labelling, storage, and manufacturer is provided in the current country-specific product information. The summary of product characteristics (SmPC) and/or leaflet provides detailed product information for investigators in the European Union and/or in other regions.
Drug: Remdesivir — Detailed information about the formulation, posology, packaging and labelling, storage, and manufacturer is provided in the current country-specific product information. The summary of product characteristics (SmPC) and/or leaflet provides detailed product information for investigators in the European Union and/or in other regions.
  Arms: Control arm
Drug: Favipiravir — Detailed information about the formulation, posology, packaging and labelling, storage, and manufacturer is provided in the current country-specific product information. The summary of product characteristics (SmPC) and/or leaflet provides detailed product information for investigators in the European Union and/or in other regions.
  Arms: Control arm

SUMMARY:
Treatment of patients hospitalised for management of moderate COVID-19 infection

DETAILED DESCRIPTION:
This is a multicentre, open-label, controlled Phase 3 study in which adults requiring hospital admission and O2 supplementation for management of moderate COVID-19 infection will be randomised in 1:1:1 to: Plitidepsin 1.5 mg arm, Plitidepsin 2.5 mg arm and Control arm

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to initiation of any study-specific procedures and study treatment.
2. Documented diagnosis of SARS-CoV-2 infection, determined by either qualitative polymerase chain reaction (PCR), antigen test by local laboratory, or any other validated method approved by the local health authority, from appropriate biological samples collected no more than 72 hours prior to study treatment on Day 1.
3. Patient meets category 5 on the 11-point WHO Clinical Progression Scale: requires hospitalisation and oxygen by mask or nasal prongs/cannula.
4. A maximum of 14 days from onset of COVID-19 symptoms to initiation of study treatment on Day 1.
5. Male or female aged ≥18 years.
6. Adequate bone marrow, liver, kidney, and metabolic function, defined by the following tests performed at local laboratory:

   * Absolute neutrophil count ≥500/mm^3 (0.5 x 10^9/L).
   * Platelet count ≥75,000/mm^3 (75 x 10^9/L).
   * Alanine transaminase (ALT), aspartate transaminase (AST) ≤3 x upper limit of normal (ULN).
   * Serum bilirubin ≤1 x ULN (or direct bilirubin <1 x ULN when total bilirubin is above ULN).
   * Calculated creatinine clearance ≥30 mL/min (Cockcroft-Gault equation).
   * Creatine phosphokinase (CPK) ≤2.5 x ULN except if the patient has had recent (i.e., in the last week) shivering episodes or trauma. In that case, the level of CPK should be ≤5 x ULN.
7. Agree not to participate in another interventional clinical trial through Day 31.
8. Females of reproductive capacity must have a negative serum or urine pregnancy test by local laboratory at study enrolment and must be non-lactating.
9. Females and males with partners of child-bearing potential must use effective contraception while on study treatment and for 6 months after last dose of plitidepsin. Patients in the control arm must use effective contraception during the time indicated in the approved product information (summary of product characteristics [SmPC] or leaflet). If no information is available in the approved product information, patients in the control arm must use effective contraception for at least one week after the study completion or the time indicated based on the investigator's discretion.

Exclusion Criteria:

1. Subjects with a pre-baseline (i.e., in the month preceding the current COVID-19 infection) impairment in general health condition for whatever reason except COVID-19, with a severe dependency for daily living activities (Barthel index ≤ 60/100) or chronic oxygen therapy.
2. Having received treatment for COVID-19 in another clinical trial in the prior 4 weeks, except documented allocation in a placebo arm.
3. Evidence of respiratory failure at the time of randomisation, based on resource utilisation requiring at least one of the following: endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula, non-invasive positive pressure ventilation, ECMO, or clinical diagnosis of respiratory failure (i.e., clinical need for one of the aforementioned therapies, which could not be administered in a resource-limited setting).
4. Patients with severe COVID-19, meeting score >5 on the 11-point WHO Clinical Progression Scale or presenting, after an initial stabilisation prior to randomisation, any of clinical signs indicative of severe systemic illness, such as respiratory rate ≥30 per minute, heart rate ≥125 per minute, or PaO2/FiO2 <300. In case a direct measure of PaO2 has not been obtained, it should be imputed according to a referenced formula. For sites located over 1000 m above sea level, PaO2/FiO2 ratio will be adjusted.
5. Patients receiving, at randomisation, treatment with antiviral therapy against SARS-CoV-2 or requiring anti-inflammatory/immunomodulating drugs beyond glucocorticoids with the exceptions listed below:

   * Prior administration of dexamethasone or equivalent glucocorticoid might be acceptable if:

     1. The total daily dose is not higher than 10 mg of dexamethasone phosphate (equivalent to dexamethasone base 8.25 mg/day) or equivalent glucocorticoids.
     2. The duration of the treatment does not exceed 72 hours prior to study treatment Day 1.
   * Prior administration of dexamethasone or equivalent glucocorticoid might be acceptable if:

     1. The total daily dose is not higher than 10 mg of dexamethasone phosphate (equivalent to dexamethasone base 8.25 mg/day) or equivalent glucocorticoids.
     2. The duration of the treatment does not exceed 72 hours prior to study treatment Day 1.
   * Prior administration of an antiviral might be acceptable in the following circumstances:

     1. For small molecules (e.g., remdesivir, molnupiravir, nirmaltrevir/ritonavir), they must have been given for an earlier stage of the disease, outside a clinical trial, and there should be a documentation of objective clinical deterioration plus evidence of persisting positivity for SARS-CoV-2 in appropriate biological samples. Last dose of previous antiviral drugs should have been administered at least 24 h before randomisation.
     2. For antiviral monoclonal antibodies, they must have been given for an earlier stage of the disease (including pre-exposure prophylaxis), outside a clinical trial, and there should be a documentation of objective clinical deterioration plus evidence of persisting positivity for SARS-CoV-2 in appropriate biological samples. Last dose of antiviral monoclonal antibodies should have been administered at least 1 week before randomisation.
6. Patients receiving treatment with chloroquine or derivatives within 8 weeks before enrolment or during the study.
7. Patients receiving treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers.
8. Viral illness (other than COVID-19) requiring therapy, except for patients with treated and adequately controlled (undetectable) human immunodeficiency virus infection.
9. Patients with uncontrolled known primary or secondary immunodeficiency, including chronic treatment with glucocorticoids (i.e., prednisone at a daily dose of >10 mg for >1 month, or another glucocorticoid at equipotent dose).
10. Any of the following cardiac conditions or risk factors:

    * Sinus bradycardia (<50 beats/min), sinus nodal dysfunction (sick sinus disease), atrioventricular block of any degree (PR >200 msec), or any other bradyarrhythmia (<50 beats/min), except for patients with permanent pacemakers;
    * Cardiac infarction, cardiac surgery or cardiac insufficiency episode within the last 6 months;
    * Known abnormal value of left ventricular ejection fraction (LVEF <low limit of normal (LLN)), unless documented confirmation of recovery (LVEF >LLN) in the previous month;
    * QT interval corrected using Fridericia's formula (QTcF) >450 msec for males or >470 msec for females;
    * History of known congenital or acquired QT prolongation;
    * Uncorrected hypokalaemia, hypocalcaemia (adjusted) and/or hypomagnesemia at screening;
    * Troponin test performed at local laboratory >1.5 x ULN; or
    * Need for an unreplaceable drug that prolongs QT and it is clearly associated with a known risk for torsades de pointes (TdP); in case of being already on treatment with these aforementioned drugs, a minimum of 4 half-lives of the drug is required before replacement (if feasible).
11. Hypersensitivity to the active ingredient or any of the excipients (mannitol, macrogolglycerol hydroxystearate, and ethanol) or patients for whom dexamethasone, antihistamine H1/H2 or antiserotoninergic agents are contraindicated.
12. Females who are pregnant (negative serum or urine pregnancy test required for all females of child-bearing potential at screening) or breast feeding.
13. Females and males with partners of child-bearing potential (females who are not surgically sterile or postmenopausal defined as amenorrhea for >12 months) who are not using at least 1 protocol specified method of contraception.
14. Any other clinically significant medical condition (including major surgery within the last 3 weeks before screening) or laboratory abnormality that, in the opinion of the investigator, would jeopardise the safety of the patient or potentially impact on patient compliance or the safety/efficacy observations in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Jimeno Doñaque, MD, PhD, Study Director — PharmaMar
Locations (28):
- Hospital Felicio Rocho, Belo Horizonte, Minas Gerais, Brazil
- "MHAT "Sveta Anna"" - Sofia AD, Sofia, Bulgaria
- Clínica de la Costa Ltda., Barranquilla, Atlántico, Colombia
- Centre Hospitalier Regional et Universitaire de Tours (CHRU Tours) - Hopital Bretonneau, Tours, France
- Greece (2):
  - Evangelismos Hospital General Hospital of Athens Evangelismos, Intensive Care Unit, Athens
  - Sotiria Hospital General Hospital of Chest Diseases of Athens "Sotiria" 3rd Department of Internal Medicine of University of Athens, Athens
- Universidad Autonoma de Nuevo Leon - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León, Mexico
- Romania (4):
  - Institutul National De Boli Infectioase "Prof. Dr. Matei Bals", Bucharest
  - Spitalul Clinic de Boli Infectioase si Tropicale Dr. Victor Babes - Bucharest, Bucharest
  - Spitalul Clinic De Boli Infectioase "Sfanta Parascheva" IASI, Sectia Boli Infectioase III, Iași
  - Spitalul Judetean de Urgenta 'Sf. Ioan cel Nou' Suceava, Sectia de Boli Infectioase, Suceava
- Spain (17):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario HM Montepríncipe, Boadilla del Monte, Madrid
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Virgen de las Nieves (HUVN), Granada
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - H. HM Sanchinarro, Madrid
  - Hospital de Emergencias Enfermera Isabel Zendal, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Instituto de Investigación Sanitaria Valdecilla (IDIVAL), Santander
  - Hospital Universitario Virgen del Rocío, Seville

REFERENCES:
- [Derived] Landete P, Caliman-Sturdza OA, Lopez-Martin JA, Preotescu L, Luca MC, Kotanidou A, Villares P, Iglesias SP, Guisado-Vasco P, Saiz-Lou EM, Del Carmen Farinas-Alvarez M, de Lucas EM, Perez-Alba E, Cisneros JM, Estrada V, Hidalgo-Tenorio C, Poulakou G, Torralba M, Fortun J, Garcia-Ocana P, Lemaignen A, Marcos-Martin M, Molina M, Paredes R, Perez-Rodriguez MT, Raev D, Ryan P, Meira F, Gomez J, Torres N, Lopez-Mendoza D, Jimeno J, Varona JF. A Phase III Randomized Controlled Trial of Plitidepsin, a Marine-Derived Compound, in Hospitalized Adults With Moderate COVID-19. Clin Infect Dis. 2024 Oct 15;79(4):910-919. doi: 10.1093/cid/ciae227. PMID 39182994

RESULTS

PARTICIPANT FLOW:
Groups:
- Plitidepsin 2.5 mg Arm: Participants received plitidepsin 2.5 mg/day intravenous (IV) in addition to dexamethasone on days 1 to 3.
- Plitidepsin 1.5 mg Arm: Participants received plitidepsin 1.5 mg/day IV in addition to dexamethasone on days 1 to 3.
- Control Arm: Participants received dexamethasone IV on Days 1 to 3. Additionally, in accordance with local treatment guidelines, participants in this group may have received a regulatory-approved antiviral treatment.
Period: Overall Study
Arm/Group | Plitidepsin 2.5 mg Arm | Plitidepsin 1.5 mg Arm | Control Arm
Started | 68 | 70 | 67
Completed | 60 | 64 | 61
Not Completed | 8 | 6 | 6
Not completed — Withdrawal by Subject | 3 | 2 | 1
Not completed — Death | 2 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Participant worsened, PI decision | 1 | 0 | 0
Not completed — Participant deterioration becoming a candidate for treatment with TZB | 1 | 0 | 0
Not completed — Participant admitted in other hospital due to a serious adverse event | 1 | 0 | 0
Not completed — Did not meet all inclusion criteria | 0 | 1 | 0
Not completed — The participant was transferred to IRCU | 0 | 1 | 0
Not completed — SAE | 0 | 1 | 0
Not completed — Discontinued as was found to be ineligible | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Plitidepsin 2.5 mg Arm | Plitidepsin 1.5 mg Arm | Control Arm | Total
Number analyzed (Participants) | 68 | 70 | 67 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (13.33) | 58.1 (14.80) | 59.3 (15.02) | 58.7 (14.34)
Age, Customized [Count of Participants; unit: Participants]
  ≥18 to 59 years | 32 | 34 | 32 | 98
  ≥60 to 64 years | 13 | 9 | 6 | 28
  ≥65 to 69 years | 8 | 11 | 11 | 30
  ≥70 to 74 years | 9 | 8 | 4 | 21
  ≥75 to 79 years | 3 | 6 | 7 | 16
  ≥80 years | 3 | 2 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 25 | 76
  Male | 43 | 44 | 42 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 35 | 21 | 89
  Not Hispanic or Latino | 35 | 35 | 46 | 116
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 63 | 62 | 64 | 189
  More than one race | 4 | 5 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Child-bearing potential, n (%) [Count of Participants; unit: Participants] — Population: Only females. Percentages were calculated based on the number of females per group as the denominator
  Participants
    Yes: number analyzed (Participants) | 25 | 26 | 25 | 76
    Yes | 4 | 5 | 4 | 13
    No, surgically sterile/post-menopausal: number analyzed (Participants) | 25 | 26 | 25 | 76
    No, surgically sterile/post-menopausal | 21 | 18 | 19 | 58
    No, other: number analyzed (Participants) | 25 | 26 | 25 | 76
    No, other | 0 | 3 | 2 | 5
Height at screening [Mean (Standard Deviation); unit: Centimeter] — Population: Height was not recorded for some participants.
  Centimeter
    number analyzed (Participants) | 66 | 67 | 65 | 198
    (all) | 167.79 (8.067) | 169.56 (8.534) | 169.25 (10.095) | 168.87 (8.921)
Weight at screening [Mean (Standard Deviation); unit: kilogram] — Population: weight was not recorded for some participants.
  kilogram
    number analyzed (Participants) | 68 | 68 | 66 | 202
    (all) | 82.72 (14.380) | 86.05 (19.778) | 87.38 (19.672) | 85.36 (18.120)
Body mass index at screening [Mean (Standard Deviation); unit: kg/m^2] — Population: not recorded for some participants
  kg/m^2
    number analyzed (Participants) | 66 | 67 | 65 | 198
    (all) | 29.45 (4.555) | 29.68 (5.617) | 30.26 (6.116) | 29.79 (5.448)
Body mass index group at screening [Count of Participants; unit: Participants]
  ≥18.5 and <25 kg/m^2 | 10 | 10 | 10 | 30
  ≥25 and <30 kg/m^2 | 31 | 35 | 26 | 92
  ≥30 and <35 kg/m^2 | 15 | 13 | 17 | 45
  ≥35 and <40 kg/m^2 | 9 | 4 | 8 | 21
  ≥40 kg/m^2 | 1 | 5 | 4 | 10
  Missing | 2 | 3 | 2 | 7
Body surface area at screening [Mean (Standard Deviation); unit: m^2] — Population: not recorded for some participants
  m^2
    number analyzed (Participants) | 66 | 67 | 65 | 198
    (all) | 1.922 (0.1787) | 1.961 (0.2252) | 1.968 (0.2299) | 1.950 (0.2123)
Periods of inclusion [Count of Participants; unit: Participants]
  Beginning of accrual - August 2021 | 2 | 1 | 2 | 5
  September 2021 - March 2022 | 56 | 55 | 51 | 162
  April 2022 - End of accrual | 10 | 14 | 14 | 38
Systolic blood pressure (mmHg) at screening [Mean (Standard Deviation); unit: mmHg] | 123.4 (18.44) | 126.9 (16.25) | 127.9 (16.24) | 126.1 (17.04)
Diastolic blood pressure (mmHg) at screening [Mean (Standard Deviation); unit: mmHg] | 74.2 (9.53) | 76.1 (9.36) | 75.0 (11.26) | 75.1 (10.05)
Pulse rate (beats/min) at screening [Mean (Standard Deviation); unit: beats/min] | 81.6 (13.72) | 83.9 (11.36) | 84.2 (13.50) | 83.2 (12.88)
Temperature (C) at screening [Mean (Standard Deviation); unit: celsius] — Population: Data not available for all participants in this cohort
  celsius
    number analyzed (Participants) | 68 | 70 | 66 | 204
    (all) | 36.91 (0.878) | 36.90 (0.899) | 36.92 (0.875) | 36.91 (0.880)
Respiration rate (breaths/min) at screening [Mean (Standard Deviation); unit: breaths/min] — Population: Data not available for all participants in this cohort
  breaths/min
    number analyzed (Participants) | 68 | 69 | 65 | 202
    (all) | 19.5 (3.49) | 19.0 (3.40) | 19.9 (3.32) | 19.4 (3.41)
Oxygen saturation (%) at screening [Mean (Standard Deviation); unit: Percentage] — Population: Data not available for all participants in this cohort
  Percentage
    number analyzed (Participants) | 68 | 69 | 67 | 204
    (all) | 96.29 (1.779) | 96.26 (1.721) | 96.44 (1.749) | 96.33 (1.743)
Fraction of inspired oxygen (%) at screening [Mean (Standard Deviation); unit: Percentage] | 26.92 (3.861) | 26.91 (3.370) | 27.94 (9.526) | 27.25 (6.191)
Vaccination status [Count of Participants; unit: Participants]
  Fully vaccinated | 35 | 36 | 32 | 103
  Non-fully vaccinated | 6 | 3 | 4 | 13
  Not vaccinated | 27 | 31 | 31 | 89
  Fully vaccinated + Non-fully vaccinated | 41 | 39 | 36 | 116
SARS-CoV-2 viral load at Day 1 [Mean (Standard Deviation); unit: log10 copies/mL] — Population: Summary was based on full analysis set
  log10 copies/mL
    number analyzed (Participants) | 47 | 56 | 55 | 158
    (all) | 5.02 (1.880) | 4.97 (1.985) | 5.06 (2.253) | 5.01 (2.040)

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Withdrawal of Supplementary Oxygen With no Subsequent Reutilisation During Remaining Study Period
Description: Time to sustained withdrawal of oxygen supplementation (in days) with no subsequent reutilisation during remaining study period is defined as the first day, from randomisation through completion of the study, on which a patient i. satisfies categories 0 to 4 on the 11-point WHO Clinical Progression Scale, and ii. has no subsequent reutilisation of oxygen supplementation (5 to 10 on the 11-point WHO Clinical Progression Scale).
  The WHO clinical progression scale provides a measure of illness severity across a range from 0 (uninfected) to 10 (dead).
Time Frame: From administration date to Day 31(±3)
Population: Intent-to-treat Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Plitidepsin 2.5 mg Arm | Plitidepsin 1.5 mg Arm | Control Arm
Number analyzed (Participants) | 68 | 70 | 67
Days | 5 [4 to 7] | 5 [4 to 6] | 7 [6 to 8]
Statistical Analysis 1: Comparison: Plitidepsin 2.5 mg Arm vs Control Arm; Plitidepsin 2.5 mg arm versus Control arm; Test type: Superiority; p = 0.8751, Log Rank — Unadjusted 2-sided p-value, for multiplicity adjustment uses the Hochberg step-up procedure; Stratified log-rank test, including the fixed effect of the treatment group and levels of the randomisation stratification factors; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.727 to 1.53] — Stratified Cox proportional-hazards regression model, including the fixed effect of the treatment group and levels of the randomisation stratification factors,
Statistical Analysis 2: Comparison: Plitidepsin 1.5 mg Arm vs Control Arm; Plitidepsin 1.5 mg arm versus Control arm; Test type: Superiority; p = 0.0625, Log Rank — Unadjusted 2-sided p-value, for multiplicity adjustment uses the Hochberg step-up procedure; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.960 to 1.96] — Stratified Cox proportional-hazards regression model, including the fixed effect of the treatment group and levels of the randomisation stratification factors

2. Secondary Outcome: Time to Sustained (i.e., With no Subsequent Readmission to Day 31) Hospital Discharge (Since Randomisation).
Description: Time to sustained (i.e., with no subsequent readmission to Day 31) hospital discharge (since randomization)
Time Frame: From administration date to Day 31(±3)
Population: Intent-to-treat Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Plitidepsin 2.5 mg Arm | Plitidepsin 1.5 mg Arm | Control Arm
Number analyzed (Participants) | 68 | 70 | 67
Days | 7 [7 to 9] | 7 [NA to NA] — NA explanation: Variability in participants with or without hospital events is insufficient to calculate the lower and upper CI | 7 [7 to 9]
Statistical Analysis 1: Comparison: Plitidepsin 2.5 mg Arm vs Control Arm; Plitidepsin 2.5 mg arm versus Control arm; Test type: Superiority; p = 0.5945, Log Rank — Unadjusted 2-sided p-value, for multiplicity adjustment uses the Hochberg step-up procedure; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.948, 95% CI 2-sided [0.655 to 1.37] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Plitidepsin 1.5 mg Arm vs Control Arm; Plitidepsin 1.5 mg arm versus Control arm; Test type: Superiority; p = 0.3358, Log Rank — Unadjusted 2-sided p-value, for multiplicity adjustment uses the Hochberg step-up procedure; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.827 to 1.70] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Clinical Status by the 11-category WHO Clinical Progression Scale on Day 8
Description: The WHO clinical progression scale provides a measure of illness severity across a range from 0 (uninfected) to 10 (dead).
  0 = Uninfected; no viral RNA detected
  1. = Ambulatory mild disease. Asymptomatic; viral RNA detected
  2. = Ambulatory mild disease. Symptomatic; independent
  3. = Ambulatory mild disease. Symptomatic; assistance needed
  4. = Hospitalized: moderate disease. Hospitalized; no oxygen therapy
  5. = Hospitalized: moderate disease. Hospitalized; oxygen by mask or nasal prongs
  6. = Hospitalized: severe diseases. Hospitalized; oxygen by NIV or high flow
  7. = Hospitalized: severe diseases. Intubation and mechanical ventilation pO2/FIO2 > 150 or SpO2/FIO2 > 200
  8. = Hospitalized: severe diseases. Mechanical ventilation pO2 /FIO2 <150 (SpO2 /FiO2 <200) or vasopressors
  9. = Hospitalized: severe diseases. Mechanical ventilation pO2 /FiO2 <150 and vasopressors, dialysis, or ECMO
  10. = dead
Time Frame: Day 8 (±1)
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Plitidepsin 2.5 mg Arm | Plitidepsin 1.5 mg Arm | Control Arm
Number analyzed (Participants) | 63 | 67 | 65
Participants
  0 = uninfected, no viral RNA detected | 6 | 10 | 3
  1 = asymptomatic, viral RNA detected | 12 | 15 | 12
  2 = symptomatic, independent | 20 | 17 | 19
  3 = symptomatic, assistance needed | 0 | 1 | 1
  4 = hospitalised, no oxygen therapy | 4 | 8 | 7
  5 = hospitalised, oxygen by mask or nasal prongs | 10 | 8 | 20
  6 = hospitalised, oxygen by NIV or high flow | 5 | 7 | 1
  7 = intubation and mechanical ventilation. pO2/FiO2 >150 or SpO2/FiO2 >200 | 4 | 1 | 2
  8 = mechanical ventilation pO2/FiO2 <150 (SpO2/FiO2 <200) or vasopressors | 1 | 0 | 0
  9 = mechanical ventilation pO2/FiO2 <150 and vasopressors, dialysis, or ECMO | 0 | 0 | 0
  10 = dead | 1 | 0 | 0
Statistical Analysis 1: Comparison: Plitidepsin 2.5 mg Arm vs Control Arm; Plitidepsin 2.5 mg arm versus Control arm; Test type: Superiority; p = 0.7252, p-value based on proportional odds model — 2-sided; Proportional odds model with fixed effects of treatment group and randomisation stratification factors; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.604 to 2.06] — Adjusted Odds Ratio and 95% CI based on a proportional odds model with fixed effects of treatment group and randomisation stratification factors
Statistical Analysis 2: Comparison: Plitidepsin 1.5 mg Arm vs Control Arm; Plitidepsin 1.5 mg arm versus Control arm; Test type: Superiority; p = 0.0910, p-value based on proportional odds model — 2-sided; Proportional odds model with fixed effects of treatment group and randomisation stratification factors; Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.920 to 3.11] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Total Duration of Advanced Oxygen Support
Description: Total duration of advanced oxygen support (high-flow nasal oxygen, extracorporeal membrane oxygenation -ECMO-, non-invasive ventilation or mechanical ventilation).
Time Frame: From administration date to Day 31(±3)
Population: Full Analysis Set; number of participants who received advanced oxygen support are presented
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Plitidepsin 2.5 mg Arm | Plitidepsin 1.5 mg Arm | Control Arm
Number analyzed (Participants) | 13 | 11 | 11
Days | 12.2 (9.71) | 10 (8.21) | 8.3 (12.66)

5. Secondary Outcome: Number of Participants in Each Study Group Requiring Admission to ICU
Description: Number of participants in each study group requiring admission to intensive care unit
Time Frame: Day 4, Day 8(±1) , Day 15(±1) and Day 31(±3)
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Plitidepsin 2.5 mg Arm | Plitidepsin 1.5 mg Arm | Control Arm
Number analyzed (Participants) | 63 | 67 | 65
participants
  From Day 1 to Day 4 | 1 [0.0402 to 8.53] | 1 [0.0378 to 8.04] | 3 [0.962 to 12.9]
  From Day 1 to Day 8 | 7 [4.59 to 21.6] | 3 [0.933 to 12.5] | 4 [1.70 to 15.0]
  From Day 1 to Day 15 | 7 [4.59 to 21.6] | 4 [1.65 to 14.6] | 4 [1.70 to 15.0]
  From Day 1 to Day 31 | 7 [4.59 to 21.6] | 5 [2.47 to 16.6] | 4 [1.70 to 15.0]

6. Secondary Outcome: Frequency of Adverse Events
Description: Adverse Event Types according to the National Cancer Institute [NCI]-Common Terminology Criteria for AEs (CTCAE v.5.0):
  The number of participants who experienced treatment-emergent adverse events (TEAEs) are presented.
Time Frame: From administration date to Day 31(±3)
Population: As Treated Population
Measure: Count of Participants; unit: Participants
Groups:
- Control Arm: Participants received dexamethasone IV on Days 1 to 3. Additionally, in accordance with local treatment guidelines, patients in this group may have received a regulatory-approved antiviral treatment.
Arm/Group | Plitidepsin 2.5 mg Arm | Plitidepsin 1.5 mg Arm | Control Arm
Number analyzed (Participants) | 63 | 67 | 65
Participants | 45 | 44 | 40

7. Secondary Outcome: Frequency of TEAEs of ≥Grade 3 According to NCI-CTCAE for Adverse Events (Version 5.0), TEAEs of Special Interest, Serious TEAEs, Serious Treatment-related TEAEs, TEAEs Leading to Treatment Discontinuation, and Deaths
Description: Frequency of treatment-emergent adverse events (TEAEs) of ≥grade 3 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 5.0), TEAEs of special interest, serious TEAEs, serious treatment-related TEAEs, TEAEs leading to treatment discontinuation, and deaths
Time Frame: From administration date to Day 31(±3)
Population: As Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Plitidepsin 2.5 mg Arm | Plitidepsin 1.5 mg Arm | Control Arm
Number analyzed (Participants) | 63 | 67 | 65
Participants
  Any TEAE Grade ≥3 | 22 | 17 | 11
  Any TEAE of special interest | 22 | 25 | 18
  Any serious TEAE | 11 | 6 | 5
  Any serious treatment-related TEAE to any study treatment | 1 | 1 | 0
  Any TEAE leading to discontinuation of any study treatment | 1 | 1 | 1
  Any TEAE leading to death | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: From Screening to Day 31 +/- 3 days
Description: As pre-specified in the approved Protocol and Statistical Analysis Plan of the study "Safety analyses will be based on the As Treated Population." Adverse events of participants not belonging to the as-treated population: One randomized participant in Plitidepsin 1.5 mg arm, that never received any study treatment, experienced an AE of adult respiratory distress syndrome.
Arm/Group | Plitidepsin 2.5 mg Arm | Plitidepsin 1.5 mg Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 2/63 | 1/67 | 2/65
Serious Adverse Events (participants affected / at risk) | 11/63 | 6/67 | 5/65
Other Adverse Events (participants affected / at risk) | 43/63 | 43/67 | 38/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plitidepsin 2.5 mg Arm (N=63) | Plitidepsin 1.5 mg Arm (N=67) | Control Arm (N=65)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (5) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plitidepsin 2.5 mg Arm (N=63) | Plitidepsin 1.5 mg Arm (N=67) | Control Arm (N=65)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (12) | 10 (10) | 4 (4)
Nausea (Gastrointestinal disorders) | 9 (9) | 8 (8) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 4 (7) | 4 (5)
Asthenia (General disorders) | 3 (3) | 3 (3) | 2 (2)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 4 (4)
Malaise (General disorders) | 0 (0) | 3 (3) | 3 (3)
Extravasation (General disorders) | 2 (2) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site phlebitis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (2)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Serum ferritin abnormal (Investigations) | 15 (18) | 13 (16) | 4 (5)
C-reactive protein increased (Investigations) | 11 (11) | 7 (11) | 5 (5)
Blood lactate dehydrogenase increased (Investigations) | 6 (6) | 6 (7) | 6 (7)
Alanine aminotransferase increased (Investigations) | 4 (4) | 7 (8) | 5 (6)
Gamma-glutamyltransferase increased (Investigations) | 5 (7) | 8 (9) | 3 (3)
Procalcitonin increased (Investigations) | 7 (7) | 4 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 3 (3) | 4 (4)
Blood glucose increased (Investigations) | 4 (4) | 4 (4) | 4 (5)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 3 (3)
Fibrin D dimer increased (Investigations) | 2 (2) | 2 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (2) | 2 (2)
Lipase increased (Investigations) | 3 (4) | 1 (1) | 0 (0)
Adjusted calcium decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0)
Oxygen saturation (Investigations) | 1 (1) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Chest X-ray abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram PR prolongation (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Interleukin level decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Interleukin level increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (14) | 12 (12) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Acquired mixed hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (8) | 7 (8) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuromyopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 7 (8) | 6 (6) | 5 (6)
Anxiety (Psychiatric disorders) | 5 (6) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Perineal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 7 (7) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 11 (11) | 9 (9) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | 2 (4)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The decision was made by the sponsor on 31 January 2023 to prematurely end the study (early termination) based on significant difficulties in the recruitment of patients, despite the implementation of corrective measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT04784559/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT04784559/SAP_001.pdf